CLINICAL TRIAL: NCT02681172
Title: Multicenter Study to Explore the Impact of Florbetaben (FBB) in Change of Diagnosis in Patients Who Are Evaluated for AD and in Whom Lumbar Puncture is Contraindicated or CSF Results Are Ambiguous
Brief Title: Impact of FBB PET Amyloid Imaging in Change of Diagnosis in Patients With AD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Piramal Imaging Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: FBB_01_02_2015; 2015-002606-37 (EudraCT Number)
Record Dates: First submitted 2016-02-04; First posted 2016-02-12 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-03

CONDITIONS: Alzheimer's Disease (AD)
Keywords: CSF; Alzheimer's Disease (AD) and related dementia; HAS recommendations
MeSH Terms: conditions — Alzheimer Disease | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neuraceq (florbetaben 18F) PET scan (Experimental): A single dose of 300 Megabecquerels (8.1 millicuries) Neuraceq will be administered per subject.
  The applied florbetaben radioactive dose will be ± 20%.
  Interventions: Drug: Neuraceq (florbetaben 18F); Procedure: PET

INTERVENTIONS:
Drug: Neuraceq (florbetaben 18F) — Florbetaben 18F is given as an i.v. injection followed by a flush of sodium chloride solution to ensure full delivery of the dose.
  Other Names: FBB
Procedure: PET — A brain PET scan is usually taken 90 minutes after the i.v. injection of florbetaben 18F.
  Other Names: Positron Emission Tomography

SUMMARY:
This phase 4 study will explore, in the context of the present French clinical practice, the impact of florbetaben 18F (FBB) in patients evaluated for AD who require a biomarker for etiologic determination of the cognitive and functional impairment, but in whom:

1. lumbar puncture was not feasible for medical conditions
2. results of cerebrospinal fluid (CSF) analysis were considered ambiguous by treating physicians
3. lumbar puncture (LP) was refused by the patient

DETAILED DESCRIPTION:
It will be conducted in an outpatient setting at the tertiary memory clinics (CMRR) in France in patients with a preliminary diagnosis based on the completion of a prior, full diagnostic workup, not more than 12 months previously - which could include, but will not be limited to brain imaging if needed (magnetic resonance imaging (MRI) or computed tomography (CT)), neuropsychological evaluation including a Mini-Mental Status Examination (MMSE), CSF examination and other examinations according to "Haute Autorité de santé" (HAS, National Authority of Health, France) Recommendations - and in whom:

1. lumbar puncture was not feasible for medical conditions
2. results of cerebrospinal fluid (CSF) analysis were considered ambiguous by treating physicians
3. lumbar puncture (LP) was refused by the patient

For all subjects the study will comprise 3 outpatient clinic visits to record information on previous work ups and to perform the FBB Positron Emission Tomography (PET) scan (Visit 1: screening/ baseline, Visit 2: PET scan, Visit 3: subject informed on the FBB PET scan result).

At Visit 1, the initial diagnosis based on previous work up will be collected and rated on a five-point Likert confidence scale by the Physician.

At Visit 2, the FBB PET scan will be performed. Adverse events will be reported during the exam and up to 7 days after the PET procedure.

At Visit 3, based on the amyloid PET scan results, change of diagnosis will be collected, in addition to physician confidence.

ELIGIBILITY:
Inclusion Criteria:

* Patients being evaluated for Alzheimer disease and related dementias according to the HAS recommendations (atypical dementia, early onset and rapid progressive dementia)
* Patients who have previously been evaluated for AD and related dementias to whom a CSF examination was recommended in the last 12 months, but lumbar puncture was contraindicated or refused or CSF results were ambiguous, or
* Patients currently being evaluated for AD and related dementias to whom a CSF examination is recommended but lumbar puncture is contraindicated or refused
* Patients have a study partner who is willing and able to accompany him/her to all clinic visits for the duration of the protocol
* Patients able to complete all clinical visits according to the protocol
* Patients able to tolerate a 20-minute FBB PET scan
* Patient or legal representative to provide informed consent for study participation, visits and data source verification.

Exclusion Criteria:

* The subject had a previous beta amyloid imaging scan
* Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol
* Is currently receiving any investigational pharmaceutical product or has participated in a clinical trial with an investigational pharmaceutical product within 30 days prior to screening and/or was administered a radiopharmaceutical within 10 radioactive half-lives prior to study drug administration in this study
* For females of childbearing age, a positive pregnancy test

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2015-10; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Ceccaldi, Prof. MD., Principal Investigator — Hôpital de La Timone, Marseille, France; Eric Guedj, Prof., Principal Investigator — Hôpital de la Timone, Marseille, France
Locations (1):
- Coordinating center (Hôpital de La Timone) and 18 associated centers in France, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ceccaldi M, Jonveaux T, Verger A, Krolak-Salmon P, Houzard C, Godefroy O, Shields T, Perrotin A, Gismondi R, Bullich S, Jovalekic A, Raffa N, Pasquier F, Semah F, Dubois B, Habert MO, Wallon D, Chastan M, Payoux P; NEUUS in AD study group; Stephens A, Guedj E. Added value of 18F-florbetaben amyloid PET in the diagnostic workup of most complex patients with dementia in France: A naturalistic study. Alzheimers Dement. 2018 Mar;14(3):293-305. doi: 10.1016/j.jalz.2017.09.009. Epub 2017 Nov 4. PMID 29107051

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase IV, multi-center study which was conducted in an outpatient setting documenting routine clinical care in the Centres Mémoire Ressources et Recherches (CMRR). Subjects were recruited in 18 active centers in France.
Groups:
- Neuraceq (Florbetaben 18F) PET Scan: A single dose of 300 Megabecquerels (8.1 millicuries) Neuraceq was administered per subject. The applied florbetaben radioactive dose was ± 20%. Neuraceq (florbetaben 18F): Florbetaben 18F was given as an i.v. injection followed by a flush of sodium chloride solution to ensure full delivery of the dose. PET: A brain PET scan was taken 90 minutes after the i.v. injection of florbetaben 18F.
Period: Overall Study
Arm/Group | Neuraceq (Florbetaben 18F) PET Scan
Started | 218
Safety Analysis Set | 205
Full Analysis Set | 205
Per Protocol Set | 205
Completed | 205
Not Completed | 13

BASELINE CHARACTERISTICS:
Population: All subjects who received any amount of florbetaben were included in the safety analysis set.
Arm/Group | Neuraceq (Florbetaben 18F) PET Scan
Number analyzed (Participants) | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102
  Male | 103

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Change of Diagnosis Comparing Pre- and Post-scan Outcomes
Description: The Physician's diagnosis was assessed before and after FBB PET scan. The initial Physician's diagnosis was collected before the PET scan, at Visit 1, based on key diagnostic results of current or previous workup. After the PET scan, the final Physician's diagnosis was collected at Visit 3, based on the amyloid PET scan results.
Time Frame: Visit 1 (baseline evaluation) and Visit 3 (up to 6 months later)
Population: All subjects who received any amount of florbetaben were included in the Safety analysis set
Measure: Count of Participants; unit: Participants
Groups:
- Safety Analysis Set: All subjects who received any amount of florbetaben were included.
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 205
Participants | 137

2. Secondary Outcome: Number of Subjects With Improved Level of Physician Confidence in Diagnosis at Visit 3
Description: The Physician's diagnostic confidence was rated on a five-point Likert scale before and after FBB PET scan. Likert scales consisted of the categories: "very weak", "weak", "moderate", "high", and "very high".
Time Frame: Visit 1 (baseline evaluation) and Visit 3 (up to 6 months later)
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 205
Participants | 167

3. Secondary Outcome: Number of Participants With a Change of Management Plan Comparing Pre- and Post-scan Outcomes
Description: For all subjects, concomitant medications were reported and any change of the management plan (e.g. new medications initiated, medications withdrawn, additional diagnostic tests ordered, referred to another specialist) was noted.
Time Frame: Visit 1 (baseline evaluation) and Visit 3 (up to 3 months later)
Population: All subjects who received any amount of florbetaben were included in the Safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 205
Participants | 164

4. Secondary Outcome: Number of Subjects With Positive FBB PET Scan
Description: PET image interpretation was performed locally in each centre by readers who had undergone training for appropriate interpretation of scans. Scans were interpreted as either "positive" or "negative" according to the approved visual assessment method.
Time Frame: Visit 3 (up to 6 months after baseline evaluation)
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 205
Participants | 132

5. Secondary Outcome: Number of Subjects With Negative FBB PET Scans
Description: as for outcome 4
Time Frame: Visit 3 (up to 6 months after baseline evaluation)
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 205
Participants | 73

6. Secondary Outcome: Number of Subjects With Contraindicated or Failed Lumbar Puncture
Description: Number of subjects with contraindicated or failed LP (anticoagulant therapy, thrombocytopenia, lumbar puncture failed, spinal problems)
Time Frame: Visit 1 (baseline evaluation)
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 205
Participants | 45

7. Secondary Outcome: Number of Subjects With Available CSF Analysis But Results Considered as Non-contributory by the Clinician
Description: Non-contributory CSF results (ambiguous CSF result, CSF result inconsistent with clinical information, uninterpretable CSF result for technical reasons)
Time Frame: Visit 1 (baseline evaluation)
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 205
Participants | 87

8. Secondary Outcome: Number of Subjects Who Refused Lumbar Puncture.
Time Frame: Visit 1 (baseline evaluation)
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 205
Participants | 75

ADVERSE EVENTS:
Time Frame: Adverse events were captured for up to 7 days after the PET scan procedure.
Arm/Group | Safety Analysis Set
All-Cause Mortality (participants affected / at risk) | 0/205
Serious Adverse Events (participants affected / at risk) | 1/205
Other Adverse Events (participants affected / at risk) | 21/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Analysis Set (N=205)
Cerebellar infarct (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Analysis Set (N=205)
Glaucoma (Eye disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Inflammation (General disorders) | 1 (1)
Injection Site Haematoma (General disorders) | 2 (2)
Injection Site Pain (General disorders) | 4 (4)
Injection Site Paraesthesia (General disorders) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Confusional State (Psychiatric disorders) | 1 (1)
Acute Kidney injury (Renal and urinary disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Cataract operation (Surgical and medical procedures) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No